CLINICAL TRIAL: NCT06511089
Title: Carotid Artery Stenting During Endovascular Treatment of Acute Ischemic Stroke: A Randomized Multicenter Clinical Trial in Patients With Acute Ischemic Stroke and Carotid Artery Stenosis Undergoing Endovascular Treatment
Brief Title: Carotid Artery Stenting During Endovascular Treatment of Acute Stroke
Acronym: CASES
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL79046.078.23
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Stroke, Acute; Stroke, Ischemic; Carotid Stenosis; Carotid Atherosclerosis; Carotid Occlusion
MeSH Terms: conditions — Stroke; Ischemic Stroke; Carotid Stenosis; Carotid Artery Diseases

STUDY DESIGN:
Masking Description: PROBE design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carotid artery stenting during endovascular thrombectomy (Experimental): In the intervention group, the cervical carotid artery lesion will be treated with a stent during the EVT (just before or directly after intracranial thrombus removal)
  Interventions: Procedure: carotid artery stenting during EVT
- No immediate carotid artery stenting during endovascular thrombectomy (Active Comparator): The control group will be treated according to the national guidelines with carotid endarterectomy of carotid artery stenting (for patients with non-disabling stroke) or medical management alone (for patients with severe disabling stroke)
  Interventions: Other: no carotid artery stenting during EVT

INTERVENTIONS:
Procedure: carotid artery stenting during EVT — Patients with an ipsilateral high grade carotid artery stenosis or occlusion of presumed atherosclerotic origin and an proximal intracranial large vessel occlusion in the anterior circulation will be randomized using a web-based randomization tool to immediate carotid artery stenting or deferred treatment strategy of carotid artery stenosis.
  In the intervention group, the cervical carotid artery lesion will be treated with a stent during the EVT (just before or directly after intracranial thrombus removal), the control group will be treated according to the national guidelines with carotid endarterectomy of carotid artery stenting (for patients with non-disabling stroke) or medical management alone (for patients with severe disabling stroke).
  Arms: Carotid artery stenting during endovascular thrombectomy
Other: no carotid artery stenting during EVT — A deferred treatment approach: carotid revascularization within two weeks after stroke onset or best medical management only, depending on the functional recovery of the patient.
  Arms: No immediate carotid artery stenting during endovascular thrombectomy

SUMMARY:
Rationale: Approximately 20% of the patients with acute ischemic stroke due to an intracranial large vessel occlusion (LVO) has a high-grade stenosis in the ipsilateral cervical carotid artery. It is uncertain whether immediate carotid artery stenting (CAS) of a cervical carotid artery stenosis during endovascular thrombectomy (EVT) is beneficial. Immediate CAS could improve cerebral perfusion and prevent recurrent ischemic stroke but could also increase the chance of intracranial hemorrhagic complications due to hyperperfusion syndrome or to the required antiplatelet treatment to prevent stent occlusion. Moreover, some patients end up with a severe disabling stroke after EVT. In these patients carotid revascularization by carotid endarterectomy (CEA) or CAS would usually not be performed but these patients would be treated by medical management only.

Objective: to assess the safety and efficacy of immediate cervical CAS during EVT in patients with acute ischemic stroke due to LVO with a high-grade stenosis >50% or occlusion of the ipsilateral cervical carotid artery.

Study design: prospective randomized open label controlled trial comparing immediate CAS during EVT versus EVT with deferred treatment of the cervical carotid artery lesion (deferred CAS/CEA or medical management alone). Outcome assessment will be blinded for treatment allocation.

DETAILED DESCRIPTION:
Background and study aims A stroke is a serious life-threatening medical condition that happens when the blood supply to part of the brain is cut off. Approximately 1 in 5 patients suffering stroke have a narrowed carotid artery. It is not yet known if early treatment to insert a tube (stent) into the narrowed artery to hold it open and prevent future stroke is worth the difficulties associated with such treatment.

Who can participate? Patients with acute ischemic stroke with a CT-angiography-proven intracranial LVO in the anterior circulation (ICA, A1, M1 or M2) as well as an ipsilateral cervical carotid artery tandem lesion of presumed atherosclerotic origin with a stenosis >50% or an ipsilateral acute proximal internal carotid artery occlusion who are treated with EVT according to the guidelines.

What does the study involve? Patients will be randomly allocated to receive either a carotid artery stent immediately after suffering a stroke, or to treatment as usual.

What are the possible benefits and risks of participating? Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All patients are being treated with EVT according to the local guidelines. The patients allocated to the intervention group will undergo CAS during EVT, which carries a risk of cerebral hyperperfusion syndrome and subsequent intracerebral hemorrhage. The potential benefits of immediate CAS during thrombectomy include: an improvement of cerebral blood flow during and after EVT. A second benefit is a lower risk of recurrent stroke in the first 14 days compared to the deferred treatment strategy. A third benefit of immediate CAS is that the patient does not need a second invasive treatment (carotid revascularization surgery (CEA or CAS) during the rehabilitation period which again carries some risk of complications. At last, the immediate CAS approach is likely to reduce health care costs.

Where is the study run from? The study will be coordinated by the University Medical Center Groningen in the Netherlands and by the University Hospital Leuven in Belgium. 26 centres (9 in Belgium and 17 in the Netherlands) will participate.

When is the study starting and how long is it expected to run for? November 2022 to November 2026

Who is funding the study? The study is part of the COllaboration of New TReatments of Acute STroke (CONTRAST) consortium (www.contrast-consortium.nl).

The study is funded by the BeNeFIT funding members (ZonMw/KCE) (the Netherlands)

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke due to proximal intracranial occlusion in the anterior circulation (intracranial ICA, M1, proximal M2) on the CT angiography
2. Stenosis >50% according to the NASCET criteria16 or initial occlusion of the ipsilateral cervical carotid artery of presumed atherosclerotic origin on baseline CT angiography
3. Eligible for EVT according to the guidelines: EVT within 6 hours of onset or EVT between 6-24 hours after onset based on perfusion CT imaging selection (conform current guidelines)
4. Baseline National Institute of Health Stroke Scale (NIHSS) score ≥2
5. Age >18 years
6. Written informed consent (deferred consent)

Exclusion Criteria:

1. Any intracranial hemorrhage
2. Cervical carotid artery stenosis or occlusion with other causes than presumed atherosclerosis (e.g. carotid artery dissection, floating thrombus, carotid web)
3. Any exclusion criterion for EVT according to the guidelines
4. Pre stroke disability (defined as a modified Rankin Scale score >2)
5. Recent gastro-intestinal or urinary tract hemorrhage (<6 weeks)
6. Recent severe head trauma (<6 weeks)
7. Recent infarction on baseline brain CT in the same vascular territory (<6 weeks)
8. Known allergy to aspirin and/or clopidogrel
9. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2026-04-05 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale score | 90 days
  Stroke-related disability measured using the Modified Rankin Scale (mRS) Score at 90 days after stroke onset.

SECONDARY OUTCOMES:
NIHSS score 24 hours | 24 hours
  Stroke severity
TICI score | during EVT
  Recanalization after EVT
Final infarct volume on brain CT scan at 24 hours | 24 hours
  Final infarct volume on brain CT scan at 24 hours
Arterial occlusive lesion score at 24 hours | 24 hours
  Arterial occlusive lesion score at 24 hours
Any stroke | 90 days
  Any ischemic, hemorrhagic stroke or TIA
Recurrent ipsilateral TIA/ischemic stroke | 90 days
  Recurrent ipsilateral TIA/ischemic stroke
Carotid re-occlusion | 24 hours and 90 days
  Carotid re-occlusion on CTA at 24 hours or duplex at 90 days
Mortality | 90 days
  Mortality
Quality of Life | 90 days
  Quality of life measured with the EQ5D-5L)

OTHER OUTCOMES:
Symptomatic Intracranial hemorrhage | 24 hours and 90 days
  Symptomatic Intracranial hemorrhage
Any intracranial hemorrhage | 24 hours and 90 days
  Any intracranial hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Uyttenboogaart, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
https://www.contrast-consortium.nl/wp-content/uploads/2021/03/SOP-publications-v1.0.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
URL: https://cases-trial.eu/

REFERENCES:
- [Derived] Maes L, Van Elk T, van der Meij A, Roelofs F, Bogaerts K, Bokkers RP, de Borst GJ, den Hertog HM, Dippel DW, Francois O, Ligot N, Lingsma HF, Majoie CB, Peluso JP, Tancredi I, van den Wijngaard IR, van der Lugt A, Yperzeele L, Zeebregts CJ, Nederkoorn PJ, Lemmens R, Uyttenboogaart M. Carotid Artery Stenting during Endovascular treatment of acute ischemic Stroke (CASES) study protocol for a multicenter randomized clinical trial. Eur Stroke J. 2025 Sep;10(3):995-1002. doi: 10.1177/23969873251319941. Epub 2025 Feb 16. PMID 39957001
- See also: trial website — https://cases-trial.eu/
- See also: Contrast Consortium — https://www.contrast-consortium.nl/